CLINICAL TRIAL: NCT05714462
Title: Effects of Beef Consumption on Skeletal Muscle Protein Homeostasis and Inflammatory Factors in Pre- and Postmenopausal Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 275449
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Menopause Related Conditions

STUDY DESIGN:
Intervention Model Description: A randomized cross-sectional controlled trial will be conducted to quantify whole-body and muscle protein turnover and skeletal muscle inflammation following 5-days of consumption of either beef or isonitrogenous plant-based sources of protein in normal/overweight and obese post-menopausal females.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- postmenopausal with normal/overweight BMI that eats primarily beef as their protein source (Experimental)
  Interventions: Other: meals consisting of primarily animal protein sources
- postmenopausal with normal/overweight BMI that eats vegetables as their protein source (Experimental)
  Interventions: Other: meals consisting of plant protein sources
- postmenopausal with obese BMI that eats primarily beef as their protein source in study meals (Experimental)
  Interventions: Other: meals consisting of primarily animal protein sources
- postmenopausal with obese BMI that eats vegetables as their protein source in study meals (Experimental)
  Interventions: Other: meals consisting of plant protein sources
- premenopausal with normal/overweight BMI that eats primarily beef as their protein source (Active Comparator)
  Interventions: Other: meals consisting of primarily animal protein sources

INTERVENTIONS:
Other: meals consisting of primarily animal protein sources — an omnivorous diet
  Arms: postmenopausal with normal/overweight BMI that eats primarily beef as their protein source; postmenopausal with obese BMI that eats primarily beef as their protein source in study meals; premenopausal with normal/overweight BMI that eats primarily beef as their protein source
Other: meals consisting of plant protein sources — an herbivorous diet
  Arms: postmenopausal with normal/overweight BMI that eats vegetables as their protein source; postmenopausal with obese BMI that eats vegetables as their protein source in study meals

SUMMARY:
This will be a randomized study to determine if animal-based protein-rich food sources can stimulate greater muscle protein turnover and whole-body protein balance and reduce skeletal muscle inflammatory markers in postmenopausal women compared to vegetarian base protein-rich foods.

DETAILED DESCRIPTION:
A randomized cross-sectional controlled trial will be conducted to quantify whole-body and muscle protein turnover and skeletal muscle inflammation following 5-days of consumption of either beef or isonitrogenous plant-based sources of protein in normal/overweight and obese post-menopausal females. A premenopausal normal/overweight group consuming beef containing study meals will also be recruited to serve as a healthy control comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women ages 50-65 (absence of menstruation for at least 12 months).
2. Premenopausal women ages 35-45 (presence of normal monthly menstruation for the past 12 months).
3. BMI of 20.0 - 34.9 kg/m2.
4. COVID-19 negative and/or asymptomatic

Exclusion Criteria:

1. Any substantial musculoskeletal injuries/diseases that have limited daily activities in the past month.
2. Unable to stop the use of anti-inflammatory drugs for the week prior to and during study.
3. Diagnosed metabolic or hormonal disease (i.e., renal, cardiovascular, thyroid, polycystic ovary syndrome, or type I/II diabetes mellitus).
4. Currently pregnant.
5. Gave birth or was lactating within previous 12 months.
6. Undergone gastric bypass/bariatric surgery.
7. Clinically significant weight gain or loss (>5% change) in the last 12 months.
8. Consuming metabolism-altering drugs or medications (i.e., corticosteroids, stimulants, insulin, thyroid medication).
9. Unable or unwilling to suspend anti-clotting medications including aspirin use for 5 days prior to Visit 4.
10. Participating in >200 minutes/week of vigorous exercise and/or >4 days/week of resistance training.
11. Unwilling to fast overnight.
12. Surgical menopause.
13. Having undergone hormone replacement therapy in the last 12 months.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Net change in muscle protein synthesis (% per day). | Study meals are eaten for 5 consecutive days.
  Change in net muscle protein synthesis between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Translational Research in Aging and Longevity, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No